CLINICAL TRIAL: NCT01209091
Title: Utility and Work Productivity Data for Economic Evaluation of Breast Cancer Therapies in the Netherlands and Sweden
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113547
Record Dates: First submitted 2010-08-30; First posted 2010-09-27 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Solid Tumours

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
Introduction: Many reimbursement authorities use economic evaluation to help guide decisions regarding the adoption of new treatments in reimbursement systems. Survival and quality of life are often the main measure of benefit used in an economic evaluation - expressed as a quality adjusted life year (QALY). In addition though, some decision makers will also consider the impact of a treatment on a patient's ability to continue working (expressed in terms of productivity). The aim of the present study is to estimate quality of life weights (utilities) and productivity loss for women with metastatic breast cancer (Human Epidermal Growth Factor Receptor 2 positive or HER 2+).

Methods: Separate surveys will be used to assess utilities and productivity in HER2+ metastatic breast cancer (MBC). To capture utilities health state descriptions or vignettes describing progressive disease, stable disease, and seven grade 3/4 adverse events (diarrhoea, fatigue, anaemia, leukopenia, anorexia, decreases in left ventricular ejection fraction (LVEF), and skin rash) will be developed. The vignettes will be developed based on a literature review and in depth interviews with women with MBC in the Netherlands and Sweden. Clinical experts in both countries will review the health states for content validity. The health states will be translated using forward and back translation. Members of the general public will rate the states (100 men and women in NL; 100 women aged 50+ in Sweden) using the visual analogue scale and Time Trade Off method to determine utility values. In a separate survey women who are currently being treated or have recently completed their treatment for MBC will be surveyed regarding the impact of disease on their ability to work using a validated work productivity measure (Work Productivity and Activity Impairment) in women in the Netherlands and Sweden.

ELIGIBILITY:
Inclusion Criteria:

Age > 18

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A hundred members of the general public will be recruited in the Netherlands and in Sweden to participate in time trade off (TTO) interviews. In Sweden in order to try to match the socio-demographic profile of women suffering from HER2+ MBC, recruitment will be aimed at females aged over 50. In the Netherlands participants will be from both genders, and of mixed age, ethnicity, education and employment status categories. In Sweden, interviews will be conducted in Stockholm, Tyresö and Malmo. In the Netherlands, interviews will be conducted in Rotterdam, Amsterdam and Colmschate.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Health utility: is a measure of strength of preference that people have for particular health states. A year in full health is arbitrarily assigned a value of 1: a state that is considered equivalent to death is assigned a value of zero

SECONDARY OUTCOMES:
Productivity loss: productive working time lost due to health related inability to work. These include the costs of lost work due to absenteeism or early retirement, impaired productivity at work, and lost or impaired leisure activity.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline